CLINICAL TRIAL: NCT01777802
Title: Observational Study of Immune Responses in Prostate, Lung, Melanoma and Breast Cancer Patients Following Stereotactic Body Radiotherapy (SBRT), Intensity Modulated Radiotherapy (IMRT) or Brachytherapy
Brief Title: Immune Responses in Prostate, Lung, Melanoma and Breast Cancer Patients Following Stereotactic Body Radiotherapy (SBRT), Intensity Modulated Radiotherapy (IMRT) or Brachytherapy
Acronym: SBRT
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 12-008383
Record Dates: First submitted 2013-01-24; First posted 2013-01-29 (Estimated); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Prostate Cancer; Breast Cancer; Lung Cancer; Melanoma
MeSH Terms: conditions — Prostatic Neoplasms; Breast Neoplasms; Lung Neoplasms; Melanoma | interventions — Brachytherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Whole Blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Prostate Cancer: Patients with prostate cancer will be treated with SBRT, IMRT or brachytherapy
  Interventions: Radiation: SBRT; Radiation: IMRT; Radiation: Brachytherapy
- Breast Cancer: Patients with breast cancer will be treated with SBRT, IMRT or brachytherapy
  Interventions: Radiation: SBRT; Radiation: IMRT; Radiation: Brachytherapy
- Lung Cancer: Patients with lung cancer will be treated with SBRT, IMRT or brachytherapy
  Interventions: Radiation: SBRT; Radiation: IMRT; Radiation: Brachytherapy
- Melanoma Cancer: Patients with melanoma cancer will be treated with SBRT, IMRT or brachytherapy
  Interventions: Radiation: SBRT; Radiation: IMRT; Radiation: Brachytherapy

INTERVENTIONS:
Radiation: SBRT
Radiation: IMRT
Radiation: Brachytherapy

SUMMARY:
Success of cancer immunotherapy is limited by the ability of solid tumors to evade local and systemic antitumoral immune responses. Several mechanisms of tumor immune evasion have been identified, including low intratumor expression of antigens and elevated expression of inhibitory co-regulatory molecules. An effective immunotherapy is one which would induce necrotic cell death and accompanying proinflammatory cytokine induction. Stereotactic Body Radiotherapy (SBRT) or Intensity Modulated Radiotherapy (IMRT) or brachytherapy, which is capable of delivering high, conformal radiation doses (>8 Gy) of tumor ablative radiation may be an effective means of conditioning a tumor bed to a state favorable to the initiation of robust antitumoral immune responses.

ELIGIBILITY:
Inclusion Criteria:

* Hormone Refractory, Metastatic Prostate Cancer, Lung Cancer, and Melanoma or Breast Cancer

Exclusion Criteria:

-Life expectancy of less than 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Oligometastatic prostate, lung, breast and melanoma patients
Sampling Method: Probability Sample
Enrollment: 98 (Actual)
Dates: Start 2013-01-02 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Change in immune biomarkers from baseline and after radiation treatments for breast, prostate, and lung cancers. | Before and after SBRT, IMRT, or brachytherapy
  Changes in baseline circulating tumor reactive immune markers after radiotherapy.

CONTACTS AND LOCATIONS:
Overall Officials: Sean S Park, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Evans JD, Morris LK, Zhang H, Cao S, Liu X, Mara KC, Stish BJ, Davis BJ, Mansfield AS, Dronca RS, Iott MJ, Kwon ED, Foote RL, Olivier KR, Dong H, Park SS. Prospective Immunophenotyping of CD8+ T Cells and Associated Clinical Outcomes of Patients With Oligometastatic Prostate Cancer Treated With Metastasis-Directed SBRT. Int J Radiat Oncol Biol Phys. 2019 Jan 1;103(1):229-240. doi: 10.1016/j.ijrobp.2018.09.001. Epub 2018 Sep 8. PMID 30205124
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials